CLINICAL TRIAL: NCT01493804
Title: Non-Invasive Study of Brain Connectivity Using Combined EEG and NIRS
Brief Title: Noninvasive Study of Brain Connectivity With EEG and NIRS
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120011; 12-CH-0011
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09-01

CONDITIONS: Healthy Volunteers
Keywords: Near Infrared Spectroscopy; EEG; Brain Connectivity; Healthy Volunteer; HV

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Different regions of the brain are activated when a person performs a task. Electroencephalograms (EEGs) and near-infrared spectroscopy (NIRS) are tests that detect changes in the brain. EEG looks at changes in electrical signals, and NIRS looks at changes in blood flow. These tests can detect local changes in brain activity in a safe and noninvasive way. Researchers want to study brain activity more closely by combining these tests.

Objectives:

- To use EEG and NIRS to study brain activity during specific tasks.

Eligibility:

- Healthy volunteers at least 18 years of age.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will have between one and five testing sessions. Each session will be 1 to 2 hours long. The tests given at each session will be determined by the researchers.
* Participants will have EEG and NIRS tests, given either separately or together. During these tests, participants will perform tasks of thinking and reasoning.
* Participants may also complete optional tests of thinking and reasoning. These tests will be given on paper or on a computer.

DETAILED DESCRIPTION:
Objective: To record near-infrared optical signal (NIRS) simultaneously with EEG signal and correlate hemodynamic and neuronal responses, and to understand brain connectivity associated with cognitive functions using combined EEG/NIRS technology

Study population: 40 healthy volunteers

Design: The study will aim to capture the dynamics of brain interactions on two different scales by combing EEG (neuronal) and NIRS (hemodynamic) techniques. We will then correlate the two responses to study the brain connectivity in a more comprehensive way.

Outcome Measures: graded changes in blood flow and blood oxygenation, measured with NIRS, along with electrical signals recorded by EEG in response to different functional tasks.

Note: This study is sponsored by the Center for Neuroscience and Regenerative Medicine (CNRM). De-identified data including imaging data sent to CNRM may be shared with outside investigators or collaborators. This data may be used for a variety of research purposes. The Henry M. Jackson Foundation for the Advancement for Military Medicine (HJF), USUHS, or DOD representatives may also access data for audit purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18 years or greater.

EXCLUSION CRITERIA:

* Healthy volunteers with any skin disease.
* Past or present hematologic abnormality of Hgb < 9.0 gm/dl.
* Healthy volunteers with any past or present vascular disease.
* Have a history of substance abuse, psychiatric, or neurological disorders
* Any medical condition that, in the opinion of the Principal Investigator, would preclude the inclusion of a patient onto this research study.
* Unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11-08; Study Completion 2017-09-01

CONTACTS AND LOCATIONS:
Overall Officials: Amir Gandjbakhche, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Akgul CB, Akin A, Sankur B. Extraction of cognitive activity-related waveforms from functional near-infrared spectroscopy signals. Med Biol Eng Comput. 2006 Nov;44(11):945-58. doi: 10.1007/s11517-006-0116-3. Epub 2006 Oct 24. PMID 17061116
- [Background] Aydore S, Mihcak MK, Ciftci K, Akin A. On temporal connectivity of PFC via Gauss-Markov modeling of fNIRS signals. IEEE Trans Biomed Eng. 2010 Mar;57(3):761-8. doi: 10.1109/TBME.2009.2020792. Epub 2009 Apr 28. PMID 19403360
- [Background] Badre D, Wagner AD. Selection, integration, and conflict monitoring; assessing the nature and generality of prefrontal cognitive control mechanisms. Neuron. 2004 Feb 5;41(3):473-87. doi: 10.1016/s0896-6273(03)00851-1. PMID 14766185